CLINICAL TRIAL: NCT04956965
Title: Frequency and Severity of Cardiac Injury in Transthyretin Cardiac Amyloidosis : an Electro Mapping Study.
Brief Title: High Resolution Three-dimensional Maps of the Right Chambers in Patient Diagnosed With Cardiac Amyloidosis
Acronym: CARTO-AMYLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: GIRCI SOHO (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19_RIPH3-03
Record Dates: First submitted 2021-06-21; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Amyloidosis; Cardiac Disease
Keywords: Cardiac amyloidosis; Transthyretin; Val122Ile; Cardiac electro-mapping; EnSite Precision
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Patient who needs electro-mapping in routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient free cardiac amyloidosis (Active Comparator): Patient with heart disease (related with rhythm disorders or conduction disorders) but free cardiac amyloidosis.
  Interventions: Radiation: Cardiac electro-mapping
- Patient with Transthyretin cardiac amyloidosis (Experimental): Patient with transthyretin cardiac amyloidosis plus heart disease (related with rhythm disorders or conduction disorders).
  Interventions: Radiation: Cardiac electro-mapping

INTERVENTIONS:
Radiation: Cardiac electro-mapping — Perform an high-resolution three-dimensional maps of cardiac electrical activity using EnSite Precision system.

SUMMARY:
Amyloid heart disease is an accumulation of fibrillar proteins in the extracellular sector of the heart.

Identified on echocardiography as Ventricular hypertrophy. The investigation of a Left Ventricular hypertrophy (LVH) is the most frequent discovery circumstance of amyloid heart disease.

Pathophysiological mechanisms poorly understood, resulting in late diagnosis. Transthyretin amyloid heart disease (CATTR) is the most common form of cardiac amyloidosis in the West Indies due to an abnormally high frequency of the Val122Ile and Val107Ile mutations of the transthyretin gene in this population. Val122Ile and Val107Ile mutated-transthyretin are the substitution of valine for isoleucine at codon 122 of the TTR gene ( V122I) and at codon 107 of the TTR gene (V107I).

Complications of CATTR are functional changes in heart cells or even death due to mechanical abnormalities (loss of contractility and increased wall stiffness cardiac arousal and conduction disturbances).

These disorders result from an electrical abnormality of the heart the reason why the cardiologist performs preventive performance of electrophysiological explorations with EnSite Precision™. It's a registration system used to detect foci of necrosis within the myocardium.

Amyloid deposits are areas devoid of electrical activity. Do they detectable by the EnSite Precision™ recording system ?

DETAILED DESCRIPTION:
Transthyretin's amyloid heart disease (CATTR) is a rare disease whose frequency is high in the Caribbean's due to a high frequency of Val122Ile, an amyloidosis prone mutation in the Transthyretin gene. The Val122Ile variant might be present in 15 to 20 000 subjects in Martinique, placing them at high risk to develop the CATTR.

CATTR results from the accumulation of amyloid deposits between the intercellular spans, resulting in mechanical cardiac abnormalities, but also in latent excitation or conduction defects: atrial and ventricular hyperexcitability, bundle branch blocks, atrio-ventricular blocks. These abnormalities require systematic electrophysiological studies and if necessary, antiarrythmic medications or pacemaker placement.

Electro-mapping of the cardiac chambers offers high-resolution three-dimensional maps of cardiac electrical activity which has been used recently to detect focal myocardial infarction.

This anatomo-functional imaging, used only once in cardiac amyloidosis, showed a correlation between areas of low voltage of the left atrial myocardium and areas of late gadolinium enhancement, a marker of amyloidosis deposit, found in cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

Controls:

* Aged 18 and more
* Have had an echocardiogram within 6 months prior to inclusion
* Have had a cardiac Holter in the 6 months prior to inclusion.
* Informed Consent given

Cases :

* Aged 18 and over
* Presence of cardiac amyloidosis with Transthyretin
* Have had an echocardiogram within 6 months prior to inclusion
* Have had a cardiac Holter monitoring in the 6 months prior to inclusion.
* Informed Consent given

Exclusion Criteria:

Controls

* Known case of amyloidosis in the immediate family
* Patient known to have amyloidosis
* Left ventricular wall thickness greater than or equal to 14 mm
* Hyperechogenicity of the left ventricular walls
* Cardiac disease which may affect electro-anatomic mapping: Right ventricular dysplasia, myocardial infarction, congenital heart disease.
* Contraindication such as pregnancy to radiological exams
* Presence of an anomaly of the vena cava
* Presence of intracavitary thrombus at cardiac echocardiography
* Patients with a pacemaker

Cases

* Cardiac disease which may affect electro-anatomic mapping: Right ventricular dysplasia, myocardial infarction, congenital heart disease.
* Contraindication such as pregnancy to radiological exams
* Presence of an anomaly of the vena cava
* Presence of intracavitary thrombus at cardiac echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of zones with abnormal electrical activity | 1 month
  Percentage of subject with at least one area of electrical inactivity (<0.1 mV) or at least one area of continuous low-voltage activity

SECONDARY OUTCOMES:
Characteristics of zones with electrical inactivity | 1 month
  Number of areas of electrical inactivity (<0.1 mV)
Zones with electrical inactivity | 1 month
  Area of surface of electrical inactivity (<0.1 mV)
Characteristics of zones with abnormal electrical activity | 1 month
  Number of areas of continuous low voltage activity
Zones with abnormal electrical activity | 1 month
  Surface of areas of continuous low voltage activity
Compare electrical activity anomaly to total longitudinal strain on cardiac ultrasound | 1 month
  Number of areas of electrical inactivity vs. total longitudinal strain on cardiac ultrasound.
Electrical activity anomaly and total longitudinal strain on cardiac ultrasound | 1 month
  Number of areas of continuous low voltage activity vs. Total longitudinal strain on cardiac ultrasound.
Compare electrical activity anomaly (surface) to total longitudinal strain on cardiac ultrasound | 1 month
  Surface of areas of electrical inactivity vs. Total longitudinal strain on cardiac ultrasound.
Electrical activity anomaly (continuous low voltage activity) and total longitudinal strain on cardiac ultrasound | 1 month
  Surface of areas of continuous low voltage activity vs. Total longitudinal strain on cardiac ultrasound.
Compare electrical activity anomaly to Brain Natriuretic Peptide (BNP) value | 1 month
  Number of areas of electrical inactivity vs. BNP value.
Electrical activity and Brain Natriuretic Peptide (BNP) value | 1 month
  Number of areas of continuous low voltage activity vs. BNP value.
Compare electrical activity anomaly (surface) to Brain Natriuretic Peptide (BNP) value | 1 month
  Surface of areas of electrical inactivity vs. BNP value.
Electrical activity anomaly (continuous low voltage activity) and Brain Natriuretic Peptide (BNP) value | 1 month
  Surface of areas of continuous low voltage activity vs. BNP value.
Compare electrical activity anomaly to the presence of severe ventricular arrhythmia | 1 month
  Number of areas of electrical inactivity vs. the presence of severe ventricular arrhythmia.
Electrical activity anomaly and presence of severe ventricular arrhythmia | 1 month
  Number of areas of continuous low voltage activity vs. the presence of severe ventricular arrhythmia.
Compare electrical activity anomaly (surface) to the presence of severe ventricular arrhythmia | 1 month
  Surface of areas of electrical inactivity vs. the presence of severe ventricular arrhythmia.
Electrical activity anomaly (continuous low voltage activity) and presence of severe ventricular arrhythmia | 1 month
  Surface of areas of continuous low voltage activity vs. the presence of severe ventricular arrhythmia.
Compare electrical activity anomaly and to the presence of an atrial arrythmia | 1 month
  Number of areas of electrical inactivity vs. the presence of an atrial fibrillation load.
Electrical activity anomaly and presence of an atrial arrythmia | 1 month
  Number of areas of continuous low voltage activity vs. the presence of an atrial fibrillation load.
Compare electrical activity anomaly (surface) to the presence of an atrial arrythmia | 1 month
  Surface of areas of electrical inactivity vs. the presence of an atrial fibrillation load.
Electrical activity anomaly (continuous low voltage activity) and presence of an atrial arrythmia | 1 month
  Surface of areas of continuous low voltage activity vs. the presence of an atrial fibrillation load.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn INAMO, MD, PhD, Study Director — CHU de Martinique; Fabrice DEMONIERE, MD, Principal Investigator — CHU de Martinique
Locations (1):
- Centre Hospitalier Universitaire de Fort-de-France, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khairy LT, Barin R, Demoniere F, Villemaire C, Billo MJ, Tardif JC, Macle L, Khairy P. Heart Rate Response in Spectators of the Montreal Canadiens Hockey Team. Can J Cardiol. 2017 Dec;33(12):1633-1638. doi: 10.1016/j.cjca.2017.08.002. Epub 2017 Oct 5. PMID 28987521
- [Result] Wilber DJ, Pappone C, Neuzil P, De Paola A, Marchlinski F, Natale A, Macle L, Daoud EG, Calkins H, Hall B, Reddy V, Augello G, Reynolds MR, Vinekar C, Liu CY, Berry SM, Berry DA; ThermoCool AF Trial Investigators. Comparison of antiarrhythmic drug therapy and radiofrequency catheter ablation in patients with paroxysmal atrial fibrillation: a randomized controlled trial. JAMA. 2010 Jan 27;303(4):333-40. doi: 10.1001/jama.2009.2029. PMID 20103757
- [Result] Parent F, Bachir D, Inamo J, Lionnet F, Driss F, Loko G, Habibi A, Bennani S, Savale L, Adnot S, Maitre B, Yaici A, Hajji L, O'Callaghan DS, Clerson P, Girot R, Galacteros F, Simonneau G. A hemodynamic study of pulmonary hypertension in sickle cell disease. N Engl J Med. 2011 Jul 7;365(1):44-53. doi: 10.1056/NEJMoa1005565. PMID 21732836
- [Result] Oliveira Da Silva L, Fabre J, Monfort A, Villeret J, Citony I, Cohen-Tenoudji P, Lebbadi M, Martin D, Molinie V, Inamo J. 'Green Apple' Heart Failure. West Indian Med J. 2014 Jul 3;63(6):673-5. doi: 10.7727/wimj.2013.255. Epub 2014 Jun 25. PMID 25803389